CLINICAL TRIAL: NCT00524849
Title: Randomized Phase 2 Study on the Relationship Between Circulating VEGF and Weekly or Every-four-week Zometa in Breast Cancer Patients With Bone Metastases
Brief Title: Zometa and Circulating Vascular Endothelial Growth Factor (VEGF) in Breast Cancer Patients With Bone Metastasis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Xichun Hu/Dr., Fudan University Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446ECN05
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Metastatic Breast Cancer; Bone Metastases
Keywords: Breast cancer; Bone metastasis; Circulating VEGF; Zoledronic acid; Angiogenesis
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional Zometa (Active Comparator): Zometa 4mg IV q4w, in combination with other antitumor agents one month after the initial dosing.
  Interventions: Drug: Zoledronic acid
- weekly Zometa (Experimental): Weekly Zometa in combination with other antitumor agents one month after the initial dosing.
  Interventions: Biological: Zoledronic acid

INTERVENTIONS:
Biological: Zoledronic acid — Zometa 1 mg weekly (intravenous)
  Other Names: Zometa
  Arms: weekly Zometa
Drug: Zoledronic acid — Zometa 4 mg every four weeks (intravenous)
  Arms: conventional Zometa

SUMMARY:
The primary objective of this study is to evaluate the effects of Zometa (zoledronic acid, 1 mg per week versus 4 mg every four weeks) on the circulating vascular endothelial growth factor (VEGF) levels in breast cancer patients with bone metastases. Sixty patients will be randomized into two groups.

DETAILED DESCRIPTION:
The administration of Zometa in short intervals has been implied to be more potent in maximizing its antitumor and antiangiogenesis effects, while dosing every four weeks is an appropriate strategy for the prevention and management of bone metastases. This study was designed to explore the relationship between dosing of Zometa and level of circulating VEGF.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Female, 18 years or older
* Histologically confirmed invasive breast cancer
* Bone metastases
* ECOG Performance Status of 0 to 2
* Life expectancy of more than 3 months
* Subject must have adequate organ function:

  * Cr ≤ 3 mg/dL (265 µmol/L)，
  * CrCl (Cockcroft & Gault) ≥ 30 mL/min，
  * Ca2+ > 8.0 mg/dL (2.0 mmol/L) and ≤ 12 mg/dL (3.0 mmol/L)
* Negative serum pregnancy test for women with childbearing potential
* Good conditions for infusion and willing to undergo phlebotomy during the whole study
* Have ceased anti-tumor treatment including chemotherapy, endocrinotherapy and bio-targeted therapy for over 28 days

Exclusion Criteria:

* Pregnant or lactating females
* History of other malignancy. However, subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Concurrent disease or condition that would make the subject inappropriate for study participation, or any serious medical disorder that would interfere with the subject's safety
* Active or uncontrolled infection
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandible); dental or fixture trauma; or a current or prior diagnosis of osteonecrosis of the jaw (ONJ); or exposed bone in the mouth; or slow healing after dental procedures
* Recent (within 6 weeks of Randomization) or planned dental or jaw surgery (e.g. extraction, implants)
* Known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure
* Concomitant with liver, brain or symptomatic lung metastases (symptoms such as hemoptysis, severe cough and shortness of breath)
* Accepted radiotherapy for solitary bone disease within 30 days before study
* Previous treatment with other bisphosphonates or radionuclides within one month before study
* Known hypersensitivity to bisphosphonates
* History of treatment with calcitonin, gallium nitrate or mithracin within 14 days before study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-11; Primary Completion 2008-08 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Circulating VEGF levels in breast cancer patients with bone metastases | one month

SECONDARY OUTCOMES:
Time to first skeletal-related event | 3 years
Time to bone progression disease | 3 years
Progression-free survival | 3 years
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Santini D, Vincenzi B, Dicuonzo G, Avvisati G, Massacesi C, Battistoni F, Gavasci M, Rocci L, Tirindelli MC, Altomare V, Tocchini M, Bonsignori M, Tonini G. Zoledronic acid induces significant and long-lasting modifications of circulating angiogenic factors in cancer patients. Clin Cancer Res. 2003 Aug 1;9(8):2893-7. PMID 12912933
- [Derived] Zhao X, Xu X, Zhang Q, Jia Z, Sun S, Zhang J, Wang B, Wang Z, Hu X. Prognostic and predictive value of clinical and biochemical factors in breast cancer patients with bone metastases receiving "metronomic" zoledronic acid. BMC Cancer. 2011 Sep 22;11:403. doi: 10.1186/1471-2407-11-403. PMID 21936956
- [Derived] Zhao X, Xu X, Guo L, Ragaz J, Guo H, Wu J, Shao Z, Zhu J, Guo X, Chen J, Zhu B, Wang Z, Hu X. Biomarker alterations with metronomic use of low-dose zoledronic acid for breast cancer patients with bone metastases and potential clinical significance. Breast Cancer Res Treat. 2010 Dec;124(3):733-43. doi: 10.1007/s10549-010-1183-6. Epub 2010 Sep 30. PMID 20882405